CLINICAL TRIAL: NCT01584037
Title: Adenovirus Vaccine Pregnancy Registry
Status: Withdrawn | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DR-501-401
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Adenovirus
Keywords: Adenovirus; Adenovirus Type 4; Adenovirus Type 7; Adenovirus Type 4 and Type 7 Vaccine, Live, Oral
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: This is a prospective, observational, exposure-registration and follow-up study of pregnant women exposed to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral and their live born offspring through the first year of life. The intent of the Adenovirus Vaccine Pregnancy Registry, Protocol DR-501-401, is to collect observational data on pregnancy outcomes, including birth defects, in women who were exposed to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral.

SUMMARY:
The primary purpose of the Adenovirus Vaccine Pregnancy Registry is to prospectively collect data concerning:

1. Pregnant women exposed to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral,
2. Potential confounding factors, and
3. The outcome of these pregnancies.

The secondary purpose of the Adenovirus Vaccine Pregnancy Registry is to evaluate the frequency of birth defects in prospectively enrolled pregnant women. This Registry is also designed to detect any unusual patterns of birth defects.

ELIGIBILITY:
Inclusion Criteria:

For women:

* U.S. Military service member, present or former
* Confirmed exposure to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral
* Received Adenovirus Type 4 and Type 7 Vaccine, Live, Oral while pregnant or has an estimated date of conception (DOC) within 6 weeks after receiving Adenovirus Type 4 and Type 7 Vaccine, Live, Oral
* Positive β-hCG test or fetal ultrasound,and
* Verbal and/or written informed consent obtained from the patient.

For live born offspring:

* Infant born to a woman meeting the above inclusion criteria and enrolled in the Registry, followed through one year post delivery, and
* Verbal and/or written informed consent obtained from the mother of the infant.

Exclusion Criteria:

* Patients who refuse to provide informed consent (verbal or written) to the Institutional Review Board (IRB)-approved informed consent.
* Females not exposed to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral within the inclusion criteria period.
* Patients not willing to meet Registry study conditions and requirements.

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will consist of:
  1. Women previously or currently enrolled in the U.S. Military who received Adenovirus Type 4 and Type 7 Vaccine, Live, Oral while pregnant or who conceived within 6 weeks of vaccine administration, and
  2. Infants born to females with confirmed exposure to Adenovirus Type 4 and Type 7 Vaccine, Live, Oral, followed through one year post delivery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Adverse Pregnancy Outcome by observation | 12 months
  Infants up to 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Vikki Brown, MD, Principal Investigator — Syneos Health
Locations (1):
- INC Research, LLC (Registry Coordinating Center), Wilmington, North Carolina, United States